CLINICAL TRIAL: NCT03847142
Title: Adapting, Scaling, and Spreading an Algorithmic Asthma Mobile Intervention to Promote Patient-Reported Outcomes Within Primary Care Settings
Brief Title: An Asthma Mobile Intervention to Promote Patient-Reported Outcomes in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-9027; R18HS025645 (AHRQ)
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Asthma
Keywords: informatics; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Through the randomized controlled trial component, there will be 2 arms, which include the ASTHMAXcel intervention and usual care delivered through the outpatient primary care setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASTHMAXcel arm (Experimental): The ASTHMAXcel arm represents the study intervention, which is a patient-facing mobile application for adult patients with asthma.
  Interventions: Other: ASTHMAXcel mobile application
- Usual care arm (Active Comparator): This arm represents usual care delivered in the outpatient primary care setting at the study sites.
  Interventions: Other: Outpatient primary care

INTERVENTIONS:
Other: ASTHMAXcel mobile application — ASTHMAXcel is a mobile application (patient-facing) that delivers guideline-based asthma education.
  Arms: ASTHMAXcel arm
Other: Outpatient primary care — Usual care delivered through the outpatient primary care setting
  Arms: Usual care arm

SUMMARY:
Through this study, the investigators will adapt the ASTHMAXcel mobile app and evaluate the adapted intervention through a randomized controlled trial.

DETAILED DESCRIPTION:
Through this study, the investigators will use patient and provider feedback to adapt the ASTHMAXcel mobile intervention, and will conduct a randomized controlled trial to test the intervention's impact on clinical and process outcomes.

ELIGIBILITY:
Inclusion Criteria:

English-speaking individuals >18 years with:

1. persistent asthma(diagnosis made by a healthcare provider) on a daily controller medication
2. able to give informed consent
3. Smartphone (iOS or Android) access

Exclusion Criteria:

1. use of oral corticosteroids in the 2 weeks prior to the baseline visit
2. pregnancy
3. severe psychiatric or cognitive problems that would prohibit an individual from completing the protocol
4. patients that previously received ASTHMAXcel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline asthma quality of life to 2, 6, and 12 months | Baseline, 2 months, 6 months, 12 months
  Patients' asthma quality of life measured by the mini-Asthma Quality of Life Questionnaire (mini-AQLQ)

SECONDARY OUTCOMES:
Patient satisfaction measured by the Client Satisfaction Questionnaire-8 | Baseline, 2 months, 6 months, 12 months
  Patient satisfaction measured by the Client Satisfaction Questionnaire-8
Provider perception of self-performance measured by the Asthma Physicians' Practice Assessment Questionnaire | Baseline, 2 months, 6 months, 12 months
  Provider perception of self-performance measured by the Asthma Physicians' Practice Assessment Questionnaire
Change from baseline asthma knowledge to 2 months, 6 months, and 12 months | Baseline, 2 months, 6 months, 12 months
  Asthma knowledge as measured by the validated KASE asthma questionnaire
Patient acceptance of ASTHMAXcel intervention as measured by the UTAUT questionnaire | Baseline, 2 months, 6 months, 12 months
  Patient acceptance of ASTHMAXcel intervention as measured by the UTAUT questionnaire
Change from baseline asthma control to 2, 6, and 12 months | Baseline, 2 months, 6 months, 12 months
  Asthma symptom burden as measured by the Asthma Control Test
Depression as measured by the Patient Health Questionnaire-9 | Baseline, 2 months, 6 months, 12 months
  Depression as measured by the Patient Health Questionnaire-9
Number of asthma emergency department visits | Baseline, 2 months, 6 months, 12 months
  Number of asthma emergency department visits
Number of asthma hospitalizations | Baseline, 2 months, 6 months, 12 months
  Number of asthma hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Sunit Jariwala, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Silverstein GD, Styke SC, Kaur S, Singh A, Green S, Jariwala SP, Feldman J. The Relationship Between Depressive Symptoms, eHealth Literacy, and Asthma Outcomes in the Context of a Mobile Health Intervention. Psychosom Med. 2023 Sep 1;85(7):605-611. doi: 10.1097/PSY.0000000000001170. Epub 2023 Jan 27. PMID 36799736